CLINICAL TRIAL: NCT03352375
Title: Can Positive Pressure Ventilation be Provided Through a Laryngeal Mask Airway in Pediatrics During Laparoscopic Inguinal Hernia Repair?
Brief Title: Positive Pressure Ventilation Through a Laryngeal Mask Airway in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Canan Tulay ISIL, Principal Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEEAH 462/17.03.2015
Record Dates: First submitted 2017-10-24; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Pediatric; Anesthesia
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: All pediatric patients, who were scheduled to undergo laparoscopic surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orotracheally Intubation (Active Comparator): Intervention:orotracheally intubation
  Interventions: Device: Orotracheally intubation
- Laryngeal Mask Airway (Active Comparator): Intervention: Laryngeal Mask Airway
  Interventions: Device: Laryngeal Mask Airway

INTERVENTIONS:
Device: Orotracheally intubation — Interventions used for airway safety and ventilation during surgical procedures
  Arms: Orotracheally Intubation
Device: Laryngeal Mask Airway — Interventions used for airway safety and ventilation during surgical procedures
  Arms: Laryngeal Mask Airway

SUMMARY:
The investigators aimed to investigate effects of intubation and laryngeal mask airway usage in pediatrics during laparoscopic inguinal hernia repair.

DETAILED DESCRIPTION:
Considering blood gas analysis, end tidal carbon dioxide measurements and airway changes, the investigators aimed to investigate effects of intubation and laryngeal mask airway usage in pediatrics during laparoscopic inguinal hernia repair in this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I, being scheduled to undergo laparoscopic inguinal hernia.

Exclusion Criteria:

* Patients, who did not want to participate, patients with severe airway deformities, patients having increased gastroesophageal regurgitation risk, reactive airway hiatal hernia, peripheric vascular disease, mental retardation, neuropsychiatric illness or an lung infection during the last 6 weeks.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
end tidal carbon dioxide | up to 200 minutes
  A parameter measured during positive pressure ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Canan Tulay Isil, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
Study data can only be shared without patients names

REFERENCES:
- [Background] Sinha A, Sharma B, Sood J. ProSeal as an alternative to endotracheal intubation in pediatric laparoscopy. Paediatr Anaesth. 2007 Apr;17(4):327-32. doi: 10.1111/j.1460-9592.2006.02127.x. PMID 17359400